CLINICAL TRIAL: NCT00936897
Title: A Randomized Open-Label Study to Evaluate the Safety and Efficacy of Denosumab and Ibandronate in Postmenopausal Women Sub-Optimally Treated With Daily or Weekly Bisphosphonates
Brief Title: A Study to Evaluate the Safety and Efficacy of Denosumab and Ibandronate in Postmenopausal Women Sub-Optimally Treated With Daily or Weekly Bisphosphonates
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20080562
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Results first posted 2012-11-29 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid; Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibandronate (Active Comparator): Ibandronate 150mg PO QM (tablet)
  Interventions: Drug: Ibandronate
- Denosumab (Experimental): denosumab 60mg Subcutaneous Q6M (pre-filled syringe)
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Ibandronate — Ibandronate 150mg PO QM (tablet)
  Arms: Ibandronate
Drug: Denosumab — denosumab 60mg SC Q6M (pre-filled syringe)
  Arms: Denosumab

SUMMARY:
This is a multi-center, randomized, open-label, parallel group, study being conducted in the United States and in Europe in postmenopausal women. Approximately 800 subjects will be randomized across about 65 sites in a 1:1 ratio to either denosumab 60mg SC Q6M, or ibandronate 150mg PO QM.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, postmenopausal women (based on medical history) 55 years or older at screening
* Postmenopause will be defined as no vaginal bleeding or spotting for at least 12 months
* If the subject is 55 - 59 years old and there is uncertainty regarding menopausal status, confirmation of serum FSH (>= 50 mIU/mL) and serum estradiol (<= 20 pg/mL) must be obtained
* If the subject is 60 years or older, evaluation of FSH and estradiol levels is not needed to confirm menopausal status
* Have received their first prescription of daily or weekly bisphosphonate therapy at least 1 month prior to screening
* May have received
* raloxifene, calcitonin, prior to initiation of daily orweekly bisphosphonate therapy.
* up to 3 doses of monthly bisphosphonate prior to initiation of daily or weekly bisphosphonate therapy
* calcium, and vitamin D
* Hormone replacement therapy (e.g. estrogen use for mitigation of menopausal symptoms)
* Subject has:
* Stopped daily or weekly bisphosphonate therapy (is denoted as non-persistent) at least one month before the screening visit, or
* Demonstrated low adherence to therapy assessed by a score of less than 6 on the OS-MMAS
* Screening BMD (g/cm2) values, at the lumbar spine OR total hip, that occur within the following ranges, based on the particular scanner that is used:

GE Lunar Lumbar spine 0.700 < or = BMD < and = 0.940 Total hip 0.504 < or = BMD < or = 0.756

Hologic Lumbar spine 0.607 < or = BMD < or = 0.827 Total hip 0.454 < or = BMD < or = 0.698 Both the initial and the repeat DXA scan of the lumbar spine OR the total hip must meet the above eligibility criteria.

* At least 2 lumbar vertebrae must be evaluable by DXA.
* At least one hip must be evaluable by DXA (eg, no history of either bilateral hip replacement or pins in both hips)
* Provide signed informed consent before any study-specific procedures are conducted

Exclusion Criteria:

* Any disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures
* Current or prior use of medications prescribed for osteoporosis treatment other than oral daily or weekly bisphosphonate
* Contraindicated to receive oral ibandronate 150mg PO QM, including
* Hypersensitivity to ibandronate 150mg PO QM or other constituents of ibandronate 150mg PO QM tablets
* Abnormalities of the esophagus, which delay esophageal emptying such as stricture or achalasia
* Inability to stand or sit upright for at least 60 minutes
* Administration of any of the following treatments within 3 months of screening
* Tibolone
* Anabolic steroids or testosterone
* Glucocorticosteroids (>= 5 mg prednisone equivalent per day for more than 10 days or a total cumulative dose of >= 50 mg)
* Vitamin D deficiency [25(OH) vitamin D level < 20 ng/mL (<49.9 nmol/L)] - Repletion will be allowed and subjects may be re-screened
* Evidence of any of the following per subject report, chart review or central laboratory result:
* Significantly impaired renal function as determined by estimated Glomerular Filtration Rate less that 30mL/min/1.73 m2 determined by the central laboratory
* Current hypo- or hypercalcemia based on the central laboratory reference ranges
* Active gastric or duodenal ulcer; or any history of significant gastrointestinal bleed requiring hospitalization or transfusion
* Known to have tested positive for human immunodeficiency virus, hepatitis C virus, or hepatitis B surface antigen
* Malignancy (except fully resected cutaneous basal cell or squamous cell carcinoma, cervical or breast ductal carcinoma in situ) within the last 5 years
* Any metabolic bone disease or secondary cause of bone loss that is not controlled and may interfere with the interpretation of the findings
* Previous participation in clinical trials with denosumab 60mg SC Q6M (regardless of treatment)
* Received any solid organ or bone marrow transplant
* Any laboratory abnormality which, in the opinion of the investigator, will prevent the subject from completing the study or interfere with the interpretation of the study results
* Known sensitivity to mammalian cell derived drug products
* Known intolerance to calcium supplements
* Currently enrolled in or has not yet completed at least 1 month since ending other investigational device or drug trial(s)
* Any physical or psychiatric disorder which, in the opinion of the investigator, will prevent the subject from completing the study or interfere with the interpretation of the study results
* Evidence of alcohol or substance-abuse within the last 12 months which the investigator believes would interfere with understanding or completing the study

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 833 (Actual)
Dates: Start 2009-07; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Miller PD, Pannacciulli N, Malouf-Sierra J, Singer A, Czerwinski E, Bone HG, Wang C, Huang S, Chines A, Lems W, Brown JP. Efficacy and safety of denosumab vs. bisphosphonates in postmenopausal women previously treated with oral bisphosphonates. Osteoporos Int. 2020 Jan;31(1):181-191. doi: 10.1007/s00198-019-05233-x. Epub 2019 Nov 28. PMID 31776637
- [Derived] Recknor C, Czerwinski E, Bone HG, Bonnick SL, Binkley N, Palacios S, Moffett A, Siddhanti S, Ferreira I, Ghelani P, Wagman RB, Hall JW, Bolognese MA, Benhamou CL. Denosumab compared with ibandronate in postmenopausal women previously treated with bisphosphonate therapy: a randomized open-label trial. Obstet Gynecol. 2013 Jun;121(6):1291-1299. doi: 10.1097/AOG.0b013e318291718c. PMID 23812464
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized from 29 July 2009 through 5 November 2010
Groups:
- Denosumab 60 mg SC Q6M: Denosumab 60 mg subcutaneous once every 6 months
- Ibandronate 150 mg PO QM: Ibandronate 150 mg oral monthly
Period: Overall Study
Arm/Group | Denosumab 60 mg SC Q6M | Ibandronate 150 mg PO QM
Started | 417 (Randomized) | 416 (Randomized)
Completed | 398 | 356
Not Completed | 19 | 60
Not completed — Withdrawal by Subject | 9 | 19
Not completed — Adverse Event | 4 | 13
Not completed — Other | 3 | 9
Not completed — Lost to Follow-up | 1 | 10
Not completed — Administrative Decision | 1 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Ineligibility Determined | 0 | 3
Not completed — Noncompliance | 0 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab 60 mg SC Q6M | Ibandronate 150 mg PO QM | Total
Number analyzed (Participants) | 417 | 416 | 833
Age Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (8.1) | 66.2 (7.8) | 66.7 (8)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 417 | 416 | 833
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 348 | 361 | 709
  Black or African American | 3 | 4 | 7
  Hispanic or Latino | 54 | 42 | 96
  Asian | 3 | 4 | 7
  American Indian or Alaska Native | 2 | 0 | 2
  Other | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Total Hip Bone Mineral Density Percent Change From Baseline at Month 12
Time Frame: Baseline to month 12
Population: All randomized subjects using regression imputation for missing post baseline data.
Measure: Mean (95% Confidence Interval); unit: Percentage Change From Baseline
Arm/Group | Denosumab 60 mg SC Q6M | Ibandronate 150 mg PO QM
Number analyzed (Participants) | 417 | 415
Percentage Change From Baseline | 2.2 [2.0 to 2.5] | 0.9 [0.6 to 1.1]
Statistical Analysis 1: Comparison: Denosumab 60 mg SC Q6M vs Ibandronate 150 mg PO QM; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 1.4, 95% CI 2-sided [1.0 to 1.8] — Denosumab - Ibandronate

2. Secondary Outcome: Serum Type-1 C-Telopeptide Percent Change From Baseline at Month 1
Time Frame: Baseline to month 1
Population: Randomized subjects who enrolled in the bone marker substudy
Measure: Median (Inter-Quartile Range); unit: Percentage Change From Baseline
Arm/Group | Denosumab 60 mg SC Q6M | Ibandronate 150 mg PO QM
Number analyzed (Participants) | 134 | 113
Percentage Change From Baseline | -81.1 [-88.0 to -70.9] | -35.0 [-51.9 to -15.3]
Statistical Analysis 1: Comparison: Denosumab 60 mg SC Q6M vs Ibandronate 150 mg PO QM; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Femoral Neck Bone Mineral Density Percent Change From Baseline at Month 12
Time Frame: Baseline to Month 12
Population: All randomized subjects using regression imputation for missing post baseline data
Measure: Mean (95% Confidence Interval); unit: Percentage Change From Baseline
Arm/Group | Denosumab 60 mg SC Q6M | Ibandronate 150 mg PO QM
Number analyzed (Participants) | 417 | 415
Percentage Change From Baseline | 1.7 [1.3 to 2.1] | 0.5 [0.1 to 0.9]
Statistical Analysis 1: Comparison: Denosumab 60 mg SC Q6M vs Ibandronate 150 mg PO QM; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 1.2, 95% CI 2-sided [0.7 to 1.7] — Denosumab - Ibandronate

4. Secondary Outcome: Lumbar Spine Bone Mineral Density Percent Change From Baseline at Month 12
Time Frame: Baseline to month 12
Population: All randomized subjects using regression imputation for missing post baseline data
Measure: Mean (95% Confidence Interval); unit: Percentage Change From Baseline
Arm/Group | Denosumab 60 mg SC Q6M | Ibandronate 150 mg PO QM
Number analyzed (Participants) | 417 | 415
Percentage Change From Baseline | 4.1 [3.7 to 4.5] | 2.1 [1.7 to 2.5]
Statistical Analysis 1: Comparison: Denosumab 60 mg SC Q6M vs Ibandronate 150 mg PO QM; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 2.0, 95% CI 2-sided [1.5 to 2.5] — Denosumab - Ibandronate

ADVERSE EVENTS:
Time Frame: 12 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events. Participant flow includes all subjects randomized to the study. Number of subjects at risk of an adverse events are based on safety population - all randomized subjects who received at least one dose of treatment.
Arm/Group | Ibandronate 150 mg PO QM | Denosumab 60 mg SC Q6M
Serious Adverse Events (participants affected / at risk) | 22/410 | 39/411
Other Adverse Events (participants affected / at risk) | 31/410 | 42/411
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate 150 mg PO QM (N=410) | Denosumab 60 mg SC Q6M (N=411)
Atrial fibrillation (Cardiac disorders) | 0 | 2
Atrioventricular block complete (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 3
Cardiac tamponade (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 2
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Femoral hernia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Internal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 3
Device failure (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Aortic injury (Injury, poisoning and procedural complications) | 1 | 0
Cardiac vein perforation (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0
Heart injury (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 1
Bladder prolapse (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aortic valve repair (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate 150 mg PO QM (N=410) | Denosumab 60 mg SC Q6M (N=411)
Upper respiratory tract infection (Infections and infestations) | 9 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.